CLINICAL TRIAL: NCT06912438
Title: Emotional Release After Trigger Point Needling to Treat Myofascial Pain of the Head and Neck - Prospective Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-25-0050-CTIL
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Dysfunction (TMD); Temporomandibular Joint and Muscle Disorder
Keywords: Myofascial Pain; Dry Needling
MeSH Terms: conditions — Temporomandibular Joint Disorders; Muscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Patients diagnosed with TMD myofascial pain which my benefit from needling and who are willing to participate would be asked to answer a series of standardized questionnaires and would be invited to 4 needling session spaced 1-2 weeks apart.
  At each injection session, all patients would be asked to fill out the "Profile of Mood States Hebrew translation" (POMS-H) questionnaire just before and just after trigger point injections. The pain using the Numerical Rating Scale (NRS) would also be recorded as well as the personal impression of improvement using a percentage scale.
  Interventions: Other: Fill out questionnaire

INTERVENTIONS:
Other: Fill out questionnaire — After signed consent all patients will be asked to fill a series of questionnaires in print. The questionnaires administered are standardized and validated in Hebrew.
  Patients will be asked to fill out:
  Diagnostic Criteria for Temporomandibular Disorders (DC-TMD) questionnaire.
  Patient Health Questionnaire 9 PHQ-9-HEB
  Emotion Regulation Questionnaire (ERQ)
  Toronto Alexithymia Scale (TAS - 20)
  At each injection session, all patients will be asked to fill out the Profile of Mood States Hebrew translation (POMS-H) before and after trigger point injections.

SUMMARY:
Temporomandibular Dysfunction (TMD) as classified by the DC-TMD has a significant psychosocial component referred to as "Axis II".

One of the methods of treatment for myofascial TMD is "needing" which could be "dry needling" using only a needle or "wet needling" using local anesthetics.

Practitioners of needling commonly observe an emotional release by the patient undergoing needling.

This study aims to record and measure the emotional state of patients just before and just after needling for myofascial TMD via questionnaires.

DETAILED DESCRIPTION:
The most common chronic pain of the orofacial region is myofascial pain related to the muscles of mastication and the neck.

Which is classified according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).

In the DC-TMD, the "Axis I" arm, namely the "physical diagnosis" includes "muscular" disorders as well as "joint" disorders.

The DC/TMD also includes the Axis II - psychosocial arm with comorbidities such as Anxiety, Depression, PTSD.

The cause of myofascial pain is poorly understood - there is no clear organic cause and the modern understanding is that most of the pain is related to processes originating in the central nervous system or specifically in the "mind" such as poor coping mechanisms, history of trauma or PTSD, anxiety, depression, as well as issues related to emotions such as emotional repression.

There are no wide consensus guidelines for the treatment of chronic myofascial pain of the masticatory muscles and various modalities are available: physiotherapy, occlusal stabilization splints, pharmacotherapy, acupuncture, biofeedback, trigger point needling, behavioral changes, psychotherapy, and hypnotherapy.

One of the most common and effective treatments of myofascial pain in general is "needling" of trigger points namely insertion of a dry needle or injection of saline, local anesthetic, or steroids into trigger points (wet needling).

This treatment is also known as "Intramuscular Stimulation" (IMS). Our department has been treating myofascial pain with trigger point injections for over 6 years. Our standard protocol is 4 separate appointments spaced 1-2 weeks apart.

Practitioners of IMS report that for many patients, shortly after needling there is a n "emotional release" expressed as change in mood, crying, recollection of memories, calmness and relaxation. This has been our experience as well.

Despite the fact that this phenomenon is well observed among practitioners - there are very few reports in the literature.

In this study, we aim to measure the qualitative dynamics of emotions following IMS as well as asses the efficacy of treatment as a product of emotional change. There would be no change in the muscles needled or the technique but rather data is collected in regards to the emotional state before and after the standard treatment.

Methods After signed consent all patients will be asked to fill a series of questionnaires in print. The questionnaires administered are standardized and validated in Hebrew.

Patients will be asked to fill out:

1. Diagnostic Criteria for Temporomandibular Disorders (DC-TMD) questionnaire.
2. Patient Health Questionnaire 9 PHQ-9-HEB
3. Emotion Regulation Questionnaire (ERQ)
4. Toronto Alexithymia Scale (TAS - 20) Clinical data will be entered in EMR (Chameleon). Patients would receive 4 appointments for treatment spaced 1 or 2 weeks apart over a period of 1-2 months.

At each injection session, all patients will be asked to fill out the Profile of Mood States Hebrew translation (POMS-H) before and after trigger point injections. The pain using the Numerical Rating Scale (NRS) would also be recorded as well as the personal impression of improvement using a percentage scale.

Patients Study patients with relevant DC/TMD axis I diagnosis who could benefit from IMS therapy would be offered a chance to join the study.

Number of participants 100 study patients

Age range 18-99

Gender Males and females

Inclusion criteria The study group will include patients which consent to the study and are diagnosed with: Myalgia/Local Myalgia or Myofascial Pain or Myofascial pain with referral or Headache attributed to TMD with or without concurrent diagnosis related to the temporomandibular joint itself.

Exclusion criteria

Patients who are not eligible for IMS therapy will be excluded:

* PLT count under 80,000
* Active or chronic infection at site of pain
* Known allergy to amide local anesthetics
* Severe bleeding disorder such as Hemophilia
* If treated with Warfarin INR over 3

Criteria for participation ceasing -

* Patient choice
* Pain is not improving after 3 sessions

Special population - excluded

* Patients under 18
* Patients with cognitive impairments unable to fully understand the questionnaires

Duration of study: 2 years

Risk for the participants:

Equivalent to risk from IMS:

* Local hematoma
* Elevated pain after injection

ELIGIBILITY:
Inclusion Criteria:

The study group will include patients which consent to the study and are diagnosed with: Myalgia/Local Myalgia or Myofascial Pain or Myofascial pain with referral or Headache attributed to TMD with or without concurrent diagnosis related to the temporomandibular joint itself.

Exclusion Criteria:

Patients who are not eligible for IMS therapy will be excluded:

* PLT count under 80,000
* Active or chronic infection at site of pain
* Known allergy to amide local anesthetics
* Severe bleeding disorder such as Hemophilia
* If treated with Warfarin INR over 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Orofacial Pain clinic at the Oral Medicine Unite - Tel Aviv Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
Shift in mood state | From enrollment to the end of the needling session (4-8 weeks)
  The researchers expect to see a shift in the mood state of patients undergoing needling.
  There are 28 domains in the POMS-H questionnaire, grouped into 5 states: Fatigue (3,12,18,23,28), Tension (1,10,19), Depression (4,8,11,15,16,21,22) and Anger (2,6,13,14,20,25), Vigor (5,7,9,17,24,26,27).
  Between the before and after of each needling session values of Fatigue, Tension, Depression, and Anger are expected to decrease and values of Vigor are expected to increase.
  This shift is expected to be seen between the beginning and the end of each needling session as well as a trend between the 1st needling session and the 4th.
Pain reducation | From enrollment to the end of the needling session (4-8 weeks)
  The researchers expect to see a decrease in pain as quantified on the Numerical Rate Scale as well as an overall improvement in pain related to baseline as depicted in percentage by the patients.

SECONDARY OUTCOMES:
Decrease in distress, anxiety, depression. | From enrollment to the end of the needling session (4-8 weeks)
  The researchers expect an improvement in rates of anxiety, depression, distress as depicted in the GAD-7, ERQ, PHQ-4, PHQ-9 questionnaire. The total value of each questionnaire is expected to decrease between the 1st and the 4th needling session.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Medicine Unite, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Needs local Helsinki Committee authorizations.

REFERENCES:
- [Background] Netz Y, Zeav A, Arnon M, Daniel S. Translating a single-word items scale with multiple subcomponents--A Hebrew translation of the Profile of Mood States. Isr J Psychiatry Relat Sci. 2005;42(4):263-70. PMID 16618060
- [Background] Haller H, Saha FJ, Ebner B, Kowoll A, Anheyer D, Dobos G, Berger B, Choi KE. Emotional release and physical symptom improvement: a qualitative analysis of self-reported outcomes and mechanisms in patients treated with neural therapy. BMC Complement Altern Med. 2018 Nov 27;18(1):311. doi: 10.1186/s12906-018-2369-4. PMID 30482194
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Fuentes-Gallardo I, Perez-Munoz M, Mayoral-Del-Moral O, Lluch-Girbes E, Prieto-Valiente L, Falla D. Effectiveness of dry needling for chronic nonspecific neck pain: a randomized, single-blinded, clinical trial. Pain. 2016 Sep;157(9):1905-1917. doi: 10.1097/j.pain.0000000000000591. PMID 27537209
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784